CLINICAL TRIAL: NCT01885533
Title: POST-RADIOIODINE GRAVES' MANAGEMENT
Brief Title: Post-Radioiodine Graves' Management: The PRAGMA-Study
Acronym: PRAGMA
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Cardiff and Vale University Health Board (Other Government); Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 110269
Record Dates: First submitted 2013-02-15; First posted 2013-06-25 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Graves' Disease
Keywords: Graves' disease; radioiodine; thyroid; hypothyroidism; Graves' orbitopathy
MeSH Terms: conditions — Graves Disease; Thyroid Diseases; Hypothyroidism; Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Post-radioiodine medication: Anti-thyroid drugs
- Post-radioiodine medications: anti-thyroid drugs and thyroxine
- Post-radiodione medication: watchful monitoring

SUMMARY:
Thyroid dysfunction following radioiodine for Graves' disease is common, potentially detrimental and avoidable. A variety of clinical strategies are employed in the post-radioiodine era util the patient is on a stable thyroid hormone replacement regimen, which include the use of anti-thyroid drugs, antithyroid drugs with thyroxine, early thyroxine replacement and watchful monitoring until the onset of hypothyroidism. Which of these is most effective in avoiding dysthyroidism, is unknown. This study aims to address this lack of evidence. It will focus on Graves' disease as this is the commonest cause of thyrotoxicosis and the commonest indication for RI therapy. It will provide an insight into potential strategies for improving important clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients 18 years of age or over, who have given written informed consent to participate in the study
* Diagnosed with Graves' disease
* Received radioiodine for treatment of Graves' disease
* Had a minimum of 12 months follow-up after RI
* Most recent RI dose 5 years ago or less at the time of enrollment

Exclusion Criteria:

* Patients unable to give informed consent
* Age 17 years or younger
* Cause of thyrotoxicosis other than Graves' disease
* Patients who have had more than one dose of radioiodine can only be included in the study once, using data pertaining to their most recent treatment episode.
* Patients who might not adequately understand verbal explanations or written information given in English, or who have special communication needs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a history of Graves' disease treated with radioiodine
Sampling Method: Probability Sample
Enrollment: 803 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of dysthyroidism post-RI between different post-RI management strategies employed by clinicians in the UK | 12 months post radio-iodine
  To compare the incidence of dysthyroidism post-RI between different post-RI management strategies employed by clinicians in the UK:
  * anti-thyroid drugs before and /or after RI
  * anti-thyroid drugs with levothyroxine before and / or after RI
  * watchful monitoring post-RI and introduction of levothyroxine when needed.

SECONDARY OUTCOMES:
Graves orbitopathy | 12 months post-radiodiodine
weight gain | 12 months
progression of Graves' orbitopathy | 12 months
patient satisfaction | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, England
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne